CLINICAL TRIAL: NCT03197129
Title: The Effect of Waiting Room's Environment on the Levels of Anxiety Experienced by Children Prior Dental Treatment
Brief Title: Waiting Room's Environment and Children Anxiety Prior Dental Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: hadasshmo
Record Dates: First submitted 2017-06-20; First posted 2017-06-23 (Actual); Results first posted 2021-11-05 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2020-02

CONDITIONS: Dental Anxiety

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SADE waiting room (Experimental): children that will wait in the SADE waiting room
  Interventions: Other: sensory adapted waiting room
- Traditional waiting room (No Intervention): children that will wait in the traditional waiting room

INTERVENTIONS:
Other: sensory adapted waiting room — The SADE waiting room: a small waiting room (2.5mx2.5m) inside the clinic with 6 seats. A lighting column that children can touch and climb on. Auditory stimuli include rhythmic music, which is heard via loudspeakers.
  Arms: SADE waiting room

SUMMARY:
The amount of time the patient has spent awaiting treatment and the nature of the waiting room environment influence the anxiety level prior treatment. The objective of the present study is to compare the effect of waiting room's environment on the levels of anxiety experienced by children, in sensory adapted dental environment (SADE) and traditional waiting rooms. A parallel randomized trial. The participants will be randomly assigned to one type of waiting room. The participants will be asked to answer Venham Picture Test (VPT) scale while waiting in the waiting room just before entering the clinic.

DETAILED DESCRIPTION:
The SADE waiting room: a small waiting room (2.5mx2.5m) inside the clinic with 6 seats. All ceiling fluorescent lighting is removed. The adapted lighting consisted of slow-moving, repetitive visual color effects created by a projector, and a lighting column that children can touch and climb on. Auditory stimuli include rhythmic music, which is heard via loudspeakers. The traditional waiting room: a waiting area outside the clinic with ten seats in one row faces the reception desk in an area of 15 square meters. The area is air-conditioned, moderately well-lit, without posters or paintings on the walls, and no reading material.

•Dental anxiety scale- Venham Picture Test (VPT) is widely used and easily administered. In this test, children are presented with eight cards, with two figures on each card, one 'anxious' figure and one 'nonanxious' figure. They are asked to choose the figure from each pair that describes how they feel at that particular time. All cards are shown in their numbered order. If an anxious figure is chosen, a score of one is recorded. If a nonanxious cartoon is chosen, a score of zero is recorded. A measure of anxiety is obtained by totaling the number of times the child picks the cartoons depicting the anxious state (minimum score, 0; maximum score, 8). The participants will be asked to answer while waiting in the waiting room just before entering the clinic.

Study design- The study is a parallel randomized trial. The participants will be randomly assigned to one type of waiting room.

Additional data- gender, age, the lengths of waiting, the purpose of the visit (examination or treatment with/without sedation), dental experience, type of waiting room, child escort.

ELIGIBILITY:
Inclusion criteria: healthy 3-10 years old boys and girls Exclusion criteria: mentally unable to understand and answer the Venham Picture Test (VPT) to assess anxiety before treatment, accepted immediately without waiting.

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 122 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-05-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Hadassah, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fux-Noy A, Zohar M, Herzog K, Shmueli A, Halperson E, Moskovitz M, Ram D. The effect of the waiting room's environment on level of anxiety experienced by children prior to dental treatment: a case control study. BMC Oral Health. 2019 Dec 30;19(1):294. doi: 10.1186/s12903-019-0995-y. PMID 31888588

RESULTS

PARTICIPANT FLOW:
Groups:
- Traditional Waiting Room: children that will wait in the traditional waiting room
  This waiting room consisted of ten seats in one row facing the reception desk, and was air-conditioned, well-lit, without posters or paintings on the walls, and no reading material.
Period: Overall Study
Arm/Group | SADE Waiting Room | Traditional Waiting Room
Started | 60 | 62
Completed | 56 | 57
Not Completed | 4 | 5
Not completed — did not answer the VPT: shyness | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SADE Waiting Room | Traditional Waiting Room | Total
Number analyzed (Participants) | 60 | 62 | 122
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Drop out
  years
    number analyzed (Participants) | 56 | 57 | 113
    (all) | 5.63 (1.87) | 5.73 (2.1) | 5.68 (1.98)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Drop out
  Participants
    number analyzed (Participants) | 56 | 57 | 113
    Female | 23 | 28 | 51
    Male | 33 | 29 | 62
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Israel | 56 | 57 | 113

OUTCOME MEASURES:

1. Primary Outcome: Dental Anxiety
Description: According to Venham Picture Test (VPT) scale. A measure of anxiety is obtained by totaling the number of times the child picks the figure depicting the anxious state :minimum score 0; maximum score 8. A score of 0 means low anxiety, a score of 8 means high anxiety.
Time Frame: Dental anxiety will be assessed while waiting in the waiting room, up to 1 hour
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SADE Waiting Room | Traditional Waiting Room
Number analyzed (Participants) | 56 | 57
units on a scale | 1.71 (2.27) | 2 (2.28)

ADVERSE EVENTS:
Time Frame: 1 year
Description: no adverse events
Arm/Group | SADE Waiting Room | Traditional Waiting Room
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/57
Other Adverse Events (participants affected / at risk) | 0/56 | 0/57

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-23): https://cdn.clinicaltrials.gov/large-docs/29/NCT03197129/Prot_SAP_000.pdf